CLINICAL TRIAL: NCT00977288
Title: A Phase IIb, Multicenter, Randomized, Placebo-Controlled, Double-Blind, Dose-Ranging Study to Assess the Efficacy and Safety of MK0859 in Japanese Patients With Dyslipidemia
Brief Title: A Study of Safety and Efficacy of MK0859 (Anacetrapib) in Japanese Patients With Dyslipidemia (0859-029)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0859-029; 2009_662
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — anacetrapib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- 1 (Experimental): MK0859 10 mg + placebo
  Interventions: Drug: anacetrapib; Drug: Comparator: Placebo
- 2 (Experimental): MK0859 40 mg + placebo
  Interventions: Drug: anacetrapib; Drug: Comparator: Placebo
- 3 (Experimental): MK0859 100 mg + placebo
  Interventions: Drug: anacetrapib; Drug: Comparator: Placebo
- 4 (Experimental): MK0859 300 mg + placebo
  Interventions: Drug: anacetrapib; Drug: Comparator: Placebo
- 5 (Experimental): MK0859 10 mg + atorvastatin 10mg
  Interventions: Drug: anacetrapib; Drug: Comparator: atorvastatin
- 6 (Experimental): MK0859 40 mg + atorvastatin 10mg
  Interventions: Drug: anacetrapib; Drug: Comparator: atorvastatin
- 7 (Experimental): MK0859 100 mg + atorvastatin 10mg
  Interventions: Drug: anacetrapib; Drug: Comparator: atorvastatin
- 8 (Experimental): MK0859 300 mg + atorvastatin 10mg
  Interventions: Drug: anacetrapib; Drug: Comparator: atorvastatin
- 9 (Placebo Comparator): Placebo + atorvastatin 10mg
  Interventions: Drug: Comparator: atorvastatin; Drug: Comparator: Placebo
- 10 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: anacetrapib — 10, 40 or 100 mg tablet of MK0859 , once daily for 8 weeks
  Other Names: MK0859
  Arms: 1; 2; 3; 4; 5; 6; 7; 8
Drug: Comparator: atorvastatin — atorvastatin tablet, 10mg, once daily for 8 weeks
  Arms: 5; 6; 7; 8; 9
Drug: Comparator: Placebo — Placebo tablet, once daily for 8 weeks
  Arms: 1; 10; 2; 3; 4; 9

SUMMARY:
This study will investigate the effect of MK0859 when administered alone and when in combination with atorvastatin in lowering Low Density Lipoprotein -Cholesterol (LDL-C) in Japanese patients with dyslipidemia.

DETAILED DESCRIPTION:
This is the dose ranging study to evaluate efficacy and safety of MK-0859 in Japanese patients.

Eligible patients were assigned to 1 of 10 treatment groups (including treatment groups with or without administrative atorvastatin) for an 8-week treatment period which was followed by a 8-week reversibility period.

As an additional follow-up, the pregnancy information from women of childbearing potential who were treated with MK-0859 in this study will be collected retrospectively for a period of 4 years after the last dose of MK-0859.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female and between the ages of 20 and 75 years diagnosed with dyslipidemia

Exclusion Criteria:

* Patients has Coronary Heart Disease (CHD) or CHD-equivalent disease (except diabetes)
* Patients has uncontrolled diabetes
* Patient is currently participating or has participated in a study with an investigational compound within the last 3 months

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The percent change from baseline in Low Density Lipoprotein -Cholesterol at week 8 | 8 weeks

SECONDARY OUTCOMES:
The percent change from baseline in High Density Lipoprotein-Cholesterol and safety (hepatitis related AEs, myalgia, rhabdomyolysis, blood pressure, laboratory tests: ALT, AST, CK, Na, Cl, bicarbonate, and K), at week 8 | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Teramoto T, Shirakawa M, Kikuchi M, Nakagomi M, Tamura S, Surks HK, McCrary Sisk C, Numaguchi H. Efficacy and safety of the cholesteryl ester transfer protein inhibitor anacetrapib in Japanese patients with dyslipidemia. Atherosclerosis. 2013 Sep;230(1):52-60. doi: 10.1016/j.atherosclerosis.2013.05.012. Epub 2013 Jun 5. PMID 23958252